CLINICAL TRIAL: NCT00248313
Title: A Randomized, Open-label Study to Compare the Safety and Efficacy of Cyclosporin Dose Reduction With Cyclosporin Elimination in de Novo Renal Allograft Recipients Receiving Rapamune
Brief Title: Study Comparing Cyclosporin Dose Reduction With Cyclosporin Elimination in Kidney Transplant Recipients Taking Sirolimus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0468E-100479
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2007-11

CONDITIONS: Kidney Disease
Keywords: Kidney Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Sirolimus

INTERVENTIONS:
Drug: Rapamune®

SUMMARY:
To assess equivalence in the rates of functional graft survival at 12 months after transplantation in patients receiving induction therapy with cyclosporin (CsA, Neoral) and Rapamune® followed by CsA dose reduction and concentration-controlled Rapamune® versus induction with CsA and Rapamune® followed by discontinuation of CsA and concentration-controlled Rapamune®.

ELIGIBILITY:
Inclusion Criteria:

* Age: = to ≥ 18 years.
* End-stage renal disease, with patients scheduled to receive a primary or secondary renal allograft from a cadaveric donor, from a living-unrelated donor, or from a living-related donor.
* Patients with second and subsequent transplants must have maintained their primary graft for at least 6 months after transplantation (with the exception of graft failure due to technical reasons).

Exclusion Criteria:

* Evidence of active systemic or localised major infection prior to initial Rapamune® administration.
* Evidence of infiltrate, cavitation, or consolidation on chest x-ray obtained during screening.
* Use of any investigational drug or treatment up to 4 weeks prior to enrolling in the study and during the 12-month treatment phase. Exception: the use of erythropoiesis stimulating products. In these cases, erythrocyte-stimulating products must be discontinued prior to administration of Rapamune®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470
Dates: Start 2000-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Kidney Function at 12 months after transplantation.

SECONDARY OUTCOMES:
Kidney function at 6 months; incidence of side effects and rejection at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer